CLINICAL TRIAL: NCT06927674
Title: Evaluation of the Global Alliance for Improved Nutrition (GAIN) DEcent LIVelihoods for Small-scale Producers Delivered Through Economic & Resilient Food Systems (DELIVER) Project in Nigeria
Brief Title: DELIVER Evaluation in Nigeria
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: Datametrics Associates Ltd (Unknown); University of Nigeria Nsukka (Other); University of Abuja (Other)
Responsible Party: Principal Investigator, Valerie Flax, Senior Research Public Health Analyst, RTI International
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 424607
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Quantity and Variety of Vegetables Consumed
Keywords: diet; vegetables; market intervention; Nigeria; agricultural production intervention; demand generation intervention
MeSH Terms: interventions — Vegetables

STUDY DESIGN:
Intervention Model Description: This evaluation will use a quasi-experimental design to assess the impact of GAIN's DELIVER program on the quantity and diversity of vegetables consumed by smallholder farmers and neighbor households. Smallholder farmers and neighbor households will be randomly selected from lists compiled by GAIN in 4 program LGAs (2 in Kano, 2 in Kaduna). The household-level impacts of the intervention will be assessed through panel surveys in intervention LGAs at baseline and endline in two groups: (1) new smallholder farmers and (2) neighbors who are not involved in the vegetable gardening project.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other)
  Interventions: Behavioral: Consumption of vegetables

INTERVENTIONS:
Behavioral: Consumption of vegetables — DELIVER is designed to address challenges of low consumption of vegetables in both variety and quantity by working with smallholder farmers to increase production and promoting healthier diets through greater vegetable consumption. The project will build the capacity of smallholder farmers in vegetable production through collaborating with lead farmers to establish demonstration plots that showcase advanced agricultural techniques and technologies. These plots will serve as training hubs for other farmers in vegetable production, postharvest handling, as well as business and market planning. DELIVER aims to increase consumption among neighbors of the smallholder farmers by asking the farmers to recruit at least one neighbor family to whom they will regularly sell vegetables. The project also includes a livelihood component that will increase market connections and access to finance for smallholder farmers.

SUMMARY:
The DEcent LIVelihoods for small-scale producers delivered through Economic & Resilient food systems in Nigeria (DELIVER) (2024-2027) project is designed to address the low per capita consumption of vegetables and variety of vegetable consumption in northern Nigeria by working with smallholder farmers to increase production and promoting healthier diets through greater vegetable consumption among farmers and their neighbors. The objective of this evaluation is to assess the effectiveness of GAIN's DELIVER program for increasing the quantity and variety of vegetables consumed by smallholder farmer households participating in the program and by neighbor households. This evaluation will use a quasi-experimental design to assess the impact of GAIN's DELIVER programs on the quantity and diversity of vegetables consumed by smallholder farmers and non-farming neighbor households. The evaluation will be guided by the RE-AIM (reach, effectiveness, adoption, implementation, maintenance) framework. RE-AIM is a framework that is useful for evaluating the program impact of multifaceted and multilevel interventions.

ELIGIBILITY:
Inclusion Criteria:

* Farmer household member or neighbor household recruited by DELIVER farmer
* Located within the intervention LGA
* Farmer must be a member who is participating in the DELIVER project
* Adult who is ≥ 18 years old
* Able to speak English or Hausa
* Provide informed consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1568 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Quantity of vegetables consumed | Baseline (April 2025), Endline (April 2027) (2 years)
  Change in the mean grams of vegetables consumed in the previous 24 hours by farmer and neighbor households
Variety of vegetables consumed | Baseline (April 2025), Endline (April 2027) (2 years)
  Change in the number of types of vegetables consumed by farmer and non-farming neighbor households

CONTACTS AND LOCATIONS:
Overall Officials: Abiodun F. Ipadeola, PhD, Principal Investigator — Datametrics Associates Ltd
Locations (1):
- Datametrics Associates Ltd., Abuja, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
Dataset will be shared through Nesstar.